CLINICAL TRIAL: NCT06912295
Title: A Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Oral Doses of HL-1186 in Healthy Participants
Brief Title: Assess the Safety, Tolerability, and Pharmacokinetics of HL-1186 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yidian Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PY-HL-1186-I-01
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HL-1186 (Experimental): Single dose ascending(SAD): participants will be randomized to receive a single dose of HL-1186 or placebo,dose ascending will be conducted sequentially from the low-dose cohort to the high-dose cohort Food effect(FE): participants will be randomized to group A or group B, to evaluate different fed conditions on the PK of HL-1186 Multiple ascending dose(MAD): participants will be randomized to receive Muliple doses of HL-1186 or placebo, dose ascending will be conducted sequentially from the low-dose cohort to the high-dose cohort
  Interventions: Drug: HL-1186
- HL-1186 placebo (Placebo Comparator): Single dose ascending(SAD): participants will be randomized to receive a single dose of HL-1186 or placebo,dose ascending will be conducted sequentially from the low-dose cohort to the high-dose cohort Food effect(FE): participants will be randomized to group A or group B, to evaluate different fed conditions on the PK of HL-1186 Multiple ascending dose(MAD): participants will be randomized to receive Muliple doses of HL-1186 or placebo, dose ascending will be conducted sequentially from the low-dose cohort to the high-dose cohort
  Interventions: Drug: HL-1186 placebo

INTERVENTIONS:
Drug: HL-1186 — HL-1186 tablet for oral administration.
  Arms: HL-1186
Drug: HL-1186 placebo — HL-1186 placebo tablet for oral administration.
  Arms: HL-1186 placebo

SUMMARY:
This single-center, randomized, double-blind, placebo-controlled, two-part study is designed to assess the safety, tolerability and PK of oral HL-1186 Tablet in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants, males and females.
2. Between the ages of 18 and 45 years old (inclusive).
3. Weighs no less than 50 kg (for males) or 45 kg (for females) and body mass index (BMI) within 19.0 to 26.0 kg/m2 (inclusive).
4. During the screening period, vital signs, physical examination, blood routine, blood biochemistry, coagulation function, urine routine, virology examination, chest X-ray, and pregnancy blood test (female) were examined, and the results did not show abnormalities or abnormalities without clinical significance.

Exclusion Criteria:

1. Females who are pregnant or breastfeeding; females/males who are prepared for having children.
2. History or presence of neurological, cardiovascular, renal, hepatic, gastrointestinal, respiratory, hematological, endocrine, or osteoarticular disorders, or any laboratory abnormalities that pose a potential danger to constitute a risk when taking the study intervention or interfere with the interpretation of data.
3. Active infectious diseases which need anti-infection treatment.
4. Significant surgery within three months and not fully recovered per investigator's judgments.
5. Significant allergies per investigator's judgments, e.g., food allergies, allergies, or atopic reactions to any components of the investigational drug or placebo, asthma attacks, etc.
6. Immunosuppressive diseases, e.g., immunodeficiency, etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-09 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of single and multiple doses of HL-1186 in healthy participants | Single ascending dose(SAD): day1 to day14; Food effect(FE): day1 to day21; Multiple ascending dose(MAD): day1 to day27
  Number of participants with adverse events, with abnormal physical examination finding, with abnormal vital signs, abnormal 12-lead electrocardiograms and abnormal laboratory tests results (hematology, urinalysis, clinical chemistry, coagulation function

SECONDARY OUTCOMES:
To assess the pharmacokinetic parameters of HL-1186 in healthy participants | Single ascending dose(SAD): day1 to day7; Food effect(FE): day1 to day14; Multiple ascending dose(MAD): day1 to day20
  Time to reach maximum concentration (Tmax)
To assess the pharmacokinetic parameters of HL-1186 in healthy participants | Single ascending dose(SAD): day1 to day7; Food effect(FE): day1 to day14; Multiple ascending dose(MAD): day1 to day20
  Maximum concentration (Cmax)
To assess the pharmacokinetic parameters of HL-1186 in healthy participants | Single ascending dose(SAD): day1 to day7; Food effect(FE): day1 to day14; Multiple ascending dose(MAD): day1 to day20
  Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration (AUC0-t)
To assess the pharmacokinetic parameters of HL-1186 in healthy participants | Single ascending dose(SAD): day1 to day7; Food effect(FE): day1 to day14; Multiple ascending dose(MAD): day1 to day20
  Elimination half time (T1/2)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangnan University Affiliated Hospital, Wuxi, China

IPD SHARING:
Plan to Share IPD: No